CLINICAL TRIAL: NCT02508298
Title: Surrogate Markers of Portal Pressure and Changes in Portal Pressure in Patients With Compensated Cirrhosis Undergoing Anti-viral Therapy
Brief Title: Surrogate Markers of Portal Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Connecticut Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GGT0037
Record Dates: First submitted 2015-01-09; First posted 2015-07-24 (Estimated); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Portal Hypertension; Cirrhosis
Keywords: ICG; ARFI; portal hypertension; cirrhosis; diagnostic study
MeSH Terms: conditions — Hypertension, Portal; Fibrosis; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Indocyanine green retention test (Active Comparator): A baseline venous sample of 5 ml of venous will be drawn for pre-infusion measurement. Under sterile conditions 0.5 mg/kg body weight of ICG will be injected into vein. Further blood samples (5 ml each) will be collected at 5, 10, 15 and 20 minute intervals after the injection from a peripheral vein in the opposite arm using another intravenous catheter. After serum is separated by centrifugation, optical densities will be measured at 804 nm using a calibrated method for measurement of ICG level s. ICG retention at 15 minutes and elimination rate constant will be calculated by fitting the serum disappearance curve to a single exponential decay equation.This will be compared to portal pressure measured by Hepatic Venous Portal Gradient (HVPG).
  Interventions: Procedure: HVPG; Drug: Indocyanine Green Retention test
- Liver stiffness measurement (Active Comparator): ARFI measurements of the liver will be obtained using a standard ultrasound probe. The patient will be lying on his back and will be asked to hold his/her breath for 2-5 seconds during measurements.These will be compared to portal pressure measured by Hepatic Venous Portal Gradient (HVPG).
  Interventions: Procedure: HVPG; Device: Liver stiffness measurement
- Spleen stiffness measurement (Active Comparator): ARFI measurements of the spleen will be obtained using a standard ultrasound probe. The patient will be lying on his back and will be asked to hold his/her breath for 2-5 seconds during measurements.These will be compared to portal pressure measured by Hepatic Venous Portal Gradient (HVPG).
  Interventions: Procedure: HVPG; Device: Spleen stiffness measurement

INTERVENTIONS:
Procedure: HVPG — HVPG will be performed by placing a placing a 7F venous catheter into a supra-hepatic vein and then advancing a 5F balloon-tipped catheter into the right hepatic vein. Wedged hepatic venous pressure (WHVP) and free hepatic venous pressure (FHVP) will be measured by connection to an external transducer and polygraph (PowerLab, ADInstruments Inc., Colorado Springs, CO). After inflating the balloon catheter, adequacy of the occlusion will be established by injection of a small amount of radiologic contrast medium. Hepatic Venous Pressure gradient (HVPG) will be calculated as the difference between WHVP and FHVP.
  Other Names: Hepatic Venous Portal Gradient
Drug: Indocyanine Green Retention test — As decribed in arm descriptions
  Other Names: ICG test
  Arms: Indocyanine green retention test
Device: Liver stiffness measurement — As decribed in arm descriptions; perfromed by ARFI
  Other Names: LS
  Arms: Liver stiffness measurement
Device: Spleen stiffness measurement — As decribed in arm descriptions; performed by ARFI
  Other Names: SS
  Arms: Spleen stiffness measurement

SUMMARY:
This is a prospective longitudinal study that will evaluate if changes (pre and post therapy) in indocyanine green (ICG) retention test and liver stiff ness (LS) and spleen stiffness (SS) as measured by acoustic radiofrequency impulse (ARFI) correlate with changes in portal pressure as determined by the hepatic vein pressure gradient (HVPG) in patients with compensated hepatitis C virus (HCV) cirrhosis undergoing antiviral therapy.

DETAILED DESCRIPTION:
Subjects will be recruited from the outpatient setting of the West Haven VA Medical Center and the Yale Liver Clinic. Subjects between 18-85 years of age with compensated cirrhosis due to chronic hepatitis C virus (HCV) infection who will be starting anti-viral therapy to treat HCV within the next 3 months will be eligible for this study. 33 subjects (assuming 10% loss to follow-up) will be recruited and their participation will last from 6-12 months. The expected duration of the study is 2 years.

The primary end point of the study is to correlate the change (from baseline to after completing anti-HCV therapy) in ICG retention test, LS and SS as measured by ARFI with HVPG. After consent has been obtained, subjects will undergo ICG retention test, ARFI imaging and HVPG measurements before and after HCV therapy. Blood samples, demographic and clinical data will be collected before and after HCV therapy. Correlations between changes in HVPG and changes in ICG, LS and SS will be assessed. With 30 patients , we will have 80% power to perform a hypothesis test of the Pearson correlation assuming an observed correlation of 0.70 and a two-sided type I error rate of 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-85
* HCV infection (HCV-RNA positive)
* Compensated cirrhosis will be defined histologically and/or clinically (presence of compatible lab findings (platelet count ≤ 150,000, total bilirubin ≥ 2, serum albumin ≤ 3.5, INR ≥ 1.2) PLUS compatible physical exam features (cutaneous stigmata, gynecomastia in men, or splenomegaly) OR compatible radiological findings (nodular liver surface, splenomegaly, and/or collaterals). (The ultimate confirmation of the diagnosis of cirrhosis will be a baseline HVPG > 5 mmHg)
* Planned anti-HCV therapy in the next 3 months

Exclusion Criteria:

* Any clinically-evident complication of cirrhosis that defines decompensation : jaundice, ascites, variceal hemorrhage, overt hepatic encephalopathy)
* Hepatocellular carcinoma
* Co-infection with HBV or HIV
* Ongoing alcohol abuse
* Occlusive portal thrombosis,
* Presence of comorbid conditions conferring a life expectancy<1 year, history of allergy to iodides, pregnancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2014-04; Primary Completion 2018-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Indocyanine Green before and after treatment of hepatitis c | 2 years
  Indocyanine Green will be obtained , this will be conducted before and after treatment for hepatitis c and is measured in mg/dl

SECONDARY OUTCOMES:
Spleen stiffness before and after treatment of hepatitis c | 2 years
  Spleen stiffness will be obtained by ARFI, this will be conducted before and after treatment for hepatitis c and is measured in m/sec
Liver stiffness before and after treatment of hepatitis c | 2 years
  Liver stiffness will be obtained by ARFI, this will be conducted before and after treatment for hepatitis c and is measured in m/sec
Hepatic venous pressure gradient before and after treatment of hepatitis c | 2 years
  Hepatic venous pressure gradient would be obtained by catheterization of the hepatic vein, this will be conducted before and after treatment for hepatitis c and is measured in mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Guadalupe Garcia-Tsao, MD, Principal Investigator — VA Connecticut Healthcare System
Locations (2):
- United States (2):
  - Yale-New Haven Hospital, New Haven, Connecticut
  - VA Connecticut Healthcare System, West Haven, Connecticut